CLINICAL TRIAL: NCT01388387
Title: Impact of Donor and Recipient CYP3A5 Genetic Polymorphism on Tacrolimus Exposure in Patients With Hepatic Transplant
Brief Title: Pharmacogenetic Study of Tacrolimus in Hepatic Transplant (CYPTAC'H)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-022488-36; CIC0203/129 (Other: Center for Clinical Research of Rennes University Hospital)
Record Dates: First submitted 2011-07-01; First posted 2011-07-06 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Hepatic Transplantation
Keywords: pharmacogenetics; pharmacokinetics; tacrolimus; genetic polymorphism; CYP3A5; liver transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tacrolimus pharmacokinetics (Experimental)
  Interventions: Other: Tacrolimus pharmacokinetics

INTERVENTIONS:
Other: Tacrolimus pharmacokinetics — tacrolimus pharmacokinetics over 12 hours

SUMMARY:
The choice of an immunosuppressant after hepatic transplant is now more difficult than before because of the increasing number of drugs available.

Pharmacokinetic, pharmacodynamic and pharmacogenetic information can help to choose the best treatment and the best dose for each patient. The genetic polymorphism of enzymes metabolizing treatments can affect their efficacy and safety. Concerning tacrolimus, CYP3A5 activity is a major determinant of the dose needed to reach target concentrations. This study is aimed at evaluating the impact of both donor and recipient CYP3A5 genetic polymorphisms on tacrolimus exposure in patients with hepatic transplant.

DETAILED DESCRIPTION:
Pharmacogenetics is a recent tool which could help to choose the best immunosuppressive therapy in patients with hepatic transplant. Indeed, the CYP3A5 gene has many polymorphisms and one of them, g.6986 A>G, is the major determinant of the variability of expression of this protein. The allele *1 (g6986A) leads to normal protein expression while the allele *3 (g.6986G) causes lack of protein expression, and their different combinations induce a great variability in tacrolimus concentrations. As cytochromes are present in the liver and intestine, in hepatic transplant, tacrolimus exposure results from both recipient (enterocytes) and donor (liver) enzymes. Recent studies demonstrated a significant role of the genotype recipient on the dose/concentration relationship and on the dose needed to reach target concentrations. However, these studies were insufficient to analyze more precisely all impacts of this polymorphism because they did not include enough patients. The purpose of the investigators study is to evaluate the impact of donor and recipient CYP3A5 genetic polymorphism on tacrolimus exposure in patients with hepatic transplant after the first administration of tacrolimus and at 7 days post transplantation, when the dose has been adapted to avoid too high blood levels and to limit serious adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years) of Caucasian origin,
* with hepatic transplant,
* who are going to be treated by tacrolimus, and
* who gave free, well-informed and written consent.

Non-inclusion Criteria:

* Participation to another protocol incompatible with the study,
* HIV patients with antiretroviral treatment,
* Patients with legal guardianship or deprived of freedom.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2012-02-22 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Exposure to tacrolimus after the first administration, using tacrolimus area under curve (AUC) between 0 and 12 hours, weighted by the dose administered. | 12 hours

SECONDARY OUTCOMES:
Pharmacokinetics after the first administration and after 7 days of treatment | 7 days
  Maximal concentration, time needed to reach maximal concentration, residual concentration 12 hours after drug administration, terminal elimination half-life, systemic clearance, AUC 0-12h/dose.
Clinical follow-up during the 3 months post transplantation | 3 months
  Prescribed tacrolimus dose, tolerance of tacrolimus (hypertension, diabetes, renal insufficiency, neurological troubles) and signs of liver rejection assessed at each follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Eric BELLISSANT, MD, PhD, Study Chair — Rennes University Hospital; Marie-Clémence VERDIER, PharmD, Study Chair — Rennes University Hospital
Locations (1):
- Service des Maladies du Foie - Hôpital de Pontchaillou, Rennes, France

REFERENCES:
- [Result] Tron C, Woillard JB, Houssel-Debry P, David V, Jezequel C, Rayar M, Balakirouchenane D, Blanchet B, Debord J, Petitcollin A, Roussel M, Verdier MC, Bellissant E, Lemaitre F. Pharmacogenetic-Whole blood and intracellular pharmacokinetic-Pharmacodynamic (PG-PK2-PD) relationship of tacrolimus in liver transplant recipients. PLoS One. 2020 Mar 12;15(3):e0230195. doi: 10.1371/journal.pone.0230195. eCollection 2020. PMID 32163483